CLINICAL TRIAL: NCT06667752
Title: A Randomized, Double Blind, Active Controlled, Parallel Group Clinical Trial to Assess the Safety and Efficacy of Nanordica Antibacterial Wound Dressing in Patients With DFUs
Brief Title: Randomized Double-Blind Trial on Safety and Efficacy of Nanordica Advanced Antibacterial Wound Dressing for Diabetic Foot Ulcer
Acronym: NM2023
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanordica Medical OU (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NM2023; CIV-ES-24-10-049337 (Other: EUDAMED)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot Infection
Keywords: DFU; Diabetic foot ulcer; Diabetic foot infection; Chronic ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Advanced Antibacterial Wound Dressing (Experimental)
  Interventions: Device: Advanced Antibacterial Wound Dressing
- Aquacel Ag+ Extra (Active Comparator)
  Interventions: Device: Aquacel Ag+ Extra

INTERVENTIONS:
Device: Advanced Antibacterial Wound Dressing — For the first 4 weeks, wound dressing will be changed twice weekly. Subsequently, dressing selection and change frequency will be managed by the investigator as part of the standard of care for another 8 weeks.
  Arms: Advanced Antibacterial Wound Dressing
Device: Aquacel Ag+ Extra — For the first 4 weeks, wound dressing will be changed twice weekly. Subsequently, dressing selection and change frequency will be managed by the investigator as part of the standard of care for another 8 weeks.
  Arms: Aquacel Ag+ Extra

SUMMARY:
This clinical trial evaluates the safety and efficacy of the Nanordica Advanced Antibacterial Wound Dressing (AAWD) in patients suffering from diabetic foot ulcers.

At least 170 participants will be randomly allocated to be treated either with AAWD or Aquacel Ag+ Extra wound dressing for a 4-week active phase (intervention) followed by an 8-week standard of care period.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written informed consent obtained prior to any study related activities.
* Males and females aged ≥18 years.
* DFU(s) present for more than 4 weeks with a maximum diameter of 4 cm.
* IWGDF/IDSA Wound infection grades 1 (absent) or 2.
* Patients willing and able to comply with scheduled visits, laboratory sampling and study procedures.
* Ankle-brachial index (ABI) 0.9-1.4 or ABI between 0.6-0.9 with ankle pressure ≥ 70 mmHg.

Exclusion Criteria:

* Ssystemic or topical antibiotic therapy within 7 days before the enrolment.
* Any wound with known associated osteomyelitis or positive probe-to-bone test.
* Previous randomization in this clinical trial.
* Surgical procedures in the same leg as the index ulcer(s) (e.g., radical debridement, ulcerectomy, skin grafting, exostectomy, amputation) within the past four weeks, or planned to during the study.
* Use of other advanced therapies directly involving the index ulcer(s) (e.g. skin substitutes, matrices, cellbased therapies or products) within the past four weeks.
* Patients suffering cardiac disorders grade NYHA IV.
* Patients suffering hepatic disorders grade Child-Pugh C.
* Stage 4 cancer.
* Women of childbearing potential who are pregnant, breast-feeding or not using adequate contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CWC at 12 weeks | 12 weeks
  complete wound closure (CWC) at 12 weeks

SECONDARY OUTCOMES:
CWC at 4 weeks | 4 weeks
  complete wound closure (CWC) at 4 weeks
Time to heal | Up to 12 weeks
  Time until complete wound closure.
Adverse events | 12 weeks
  Number and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (11):
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn, Harju
  - North Estonia Medical Centre Foundation, Tallinn, Harju
  - Tartu University Hospital, Tartu, Tartu
- Spain (8):
  - Centro de Salud de Arcos de la Frontera, Arcos de la Frontera, Cádiz
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Centro de Salud San Benito, Jerez de la Frontera, Cádiz
  - Hospital de León, León, León
  - Clínica Universitaria de Podología de la Universidad Complutense de Madrid, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario de Donostia, San Sebastián

IPD SHARING:
Plan to Share IPD: Undecided